CLINICAL TRIAL: NCT01317888
Title: An Access Protocol for Continued Use of Anti-Epidermal Growth Factor Receptor-425 (Anti-EGFr-425) Monoclonal Antibody Radiolabeled With 1-125 for High Grade Gliomas
Brief Title: Access Protocol for MAB-425 Radiolabeled With I-125 for High Grade Gliomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Drexel University (Other)
Responsible Party: Luther W. Brady, M.D., Drexel University College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18508; 1043323 (Other: Drexel University College of Medicine IRB)
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-01

CONDITIONS: Glioblastoma Multiforme; Astrocytoma Anaplastic Foci
Keywords: high grade gliomas of the brain; anti-body treatment; survival
MeSH Terms: conditions — Glioblastoma | interventions — Iodine-125

ARMS (1):
- Treated with MAB-425 (Experimental): All patients receive the same treatment of MAb-425 +Iodine 125 in a total of three injections.
  Interventions: Drug: MAB-425 radiolabeled with I-125

INTERVENTIONS:
Drug: MAB-425 radiolabeled with I-125 — MAb425 anti-epidermal growth receptor) and Iodine-125 will be given as an injection for a total of three treatments each separated by one week.

SUMMARY:
The purpose of this access protocol is to allow patients with brain tumors who had previously received 125I-MAB 425 to receive additional course(s) of 125I-MAB 425 until their brain tumor begins to grow, they develop side effects to the treatment, or their medical condition changes (e.g., you become pregnant, become infected with human immunodeficiency virus (HIV) or develop another cancer).

ELIGIBILITY:
Inclusion Criteria:

* 18 Years or Older
* Previous treatment with at least one course of 125I-MAB 425 (one course = 3 infusions)
* Karnofsky performance status > 70%
* Hemoglobin > 10.0 g/dL, White Blood Cells > 4,000/mm3, Platelets > 100,000/mm3, BUN < 25 mg/dL, Creatinine < 1.5 mg/dL
* Signed informed consent
* Pathologic confirmation of GBM or AAF
* A negative beta hCG test for women of childbearing potential
* Negative HAMA test

Exclusion Criteria:

* Metastases or Second Primary Cancer
* Iodine allergy
* Inability to tolerate oral intake of Lugol's solution
* HIV Infection
* Positive HAMA test
* Pregnancy
* Uncontrolled Seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of disease progression | 3 months after first course with follow-up
  For the treatment to not have failed, diagnostic scans (enhanced MRI's and/or CT scans) must show nothing greater than or equal to a 25% increase in the sum of the area of the tumor measurements from baseline